CLINICAL TRIAL: NCT02869269
Title: A Study of Circulating Immune Cell Activity Changes in Blood of Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Associate professor, Konkuk University Medical Center
Other Study IDs: KUH1160096
Record Dates: First submitted 2016-07-15; First posted 2016-08-16 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early stage: patients who diagnosed as TNM stage 1 and 2
  Interventions: Device: Early stage
- Late stage: patients who diagnosed as TNM stage 3 and 4
  Interventions: Device: Late stage

INTERVENTIONS:
Device: Early stage — patients who classed as clinical stage 1 and 2
  Other Names: stage1+2
  Groups: Early stage
Device: Late stage — patients who classed as clinical stage 3 and 4
  Other Names: stage3+4
  Groups: Late stage

SUMMARY:
Previous studies have shown that colorectal cancer patients' prognosis and overall survival was related with immune cell expression in patients' tissue. However, the circulating immune cell activity changes in patients' blood has few studies. The purpose of this study is to analyze the variation of circulating immune cell activity in colorectal patients' blood which is classed as clinical staging.

DETAILED DESCRIPTION:
The patients were classed as clinical staging

1. Early (stage1+2) and Late(stage3+4)
2. regional lymph node metastasis
3. Distant metastasis
4. TNM stage

ELIGIBILITY:
Inclusion Criteria:

* patient who was planned to undergo colorectal cancer surgery.

Exclusion Criteria:

* age < 20 years old
* history of hypersensitivity reaction in propofol or sevoflurane
* history of previous cancer
* patient with ongoing inflammation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal surgery
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Circulating helper T cell activity | preoperative time
  change of expression level of T cell (0~100 %)

SECONDARY OUTCOMES:
Cytotoxic T cell and natural killer cell activity | preoperative time
  change of expression level Cytotoxic T cell and natural killer cell(0~100 %)from 0 to 100)

OTHER OUTCOMES:
CD4 and Treg cell activity and change of percentage of CD39 and CD73 | preoperative time
  change of expression level of CD4 and Treg cell activity and change of percentage of CD39 and CD73(0~100 %)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D,Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No